CLINICAL TRIAL: NCT03961425
Title: Cardia Carbonaid VS Standard Cannula VS NO CO2 Approach: Impact on Time to Complete Deairing and Clinical Neurological Events; a Randomized Prospective Study.
Brief Title: CO2 Field Saturating Alternative Techniques Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Principal Investigator, Luca Weltert, Professor of Biostatistics, Heart Surgeon, Cardiochirurgia E.H.
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-01
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Embolism Air Post-Procedural

STUDY DESIGN:
Intervention Model Description: Random allocation in 1:1:1 to either NO CO2, CO2 with non specific cannula, CO2 with dedicated diffuser
Who Masked: Outcomes Assessor
Masking Description: Clinical Outcomes are assessed by ICU physicians and the intraoperative strategy is not disclosed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NO CO2 (Active Comparator): Traditional De Airing maneuver
  Interventions: Behavioral: NO CO2
- CO2 Cannula (Active Comparator): CO2 at 8 l/min since 2 minutes before aortic cross clamp delivered by non specific needle cannula
  Interventions: Device: CO2 Cannula
- CO2 Cardia (Active Comparator): CO2 at 8 l/min since 2 minutes before aortic cross clamp delivered by commercial diffuser Cardia
  Interventions: Device: CO2 Cardia

INTERVENTIONS:
Behavioral: NO CO2 — Traditional mechanical Deairing
  Arms: NO CO2
Device: CO2 Cannula — NON specific, low cost delivery system
  Other Names: NON specific, low cost delivery system
  Arms: CO2 Cannula
Device: CO2 Cardia — Specific Commercial CO2 Diffuser
  Other Names: Specific Commercial CO2 Diffuser
  Arms: CO2 Cardia

SUMMARY:
Prospective Randomized study comparing three strategy of deairing (NO CO2 insufflation, CO2 insufflation with non specific cannula, CO2 insufflation with commercial dedicated diffuser) as regarding Time to Complete Deairing measured from declamping via TEE Echo and Neurological Events at Wake Up

DETAILED DESCRIPTION:
The impact of air bubbles into the cerebral circulation after open heart surgery has been a topic of discussion since the introduction of the heart-lung machine, and flooding the surgical field with CO2, which is heavier than Azote and Oxygen but over ten times more soluble seems a promising technique to minimize the presence of air microemboli. However very few studies have been conducted to ascertain what is the most efficient way to administer this treatment, or even of this treatment really impacts deairing time and clinical neurological events.

This study aims at comparing the use of CO2 (administered in two different ways: a simple cannula, which might be prone to emulsioning air and CO2 not reaching a complete CO2 saturation and a specific commercial diffuser which states promises complete filed saturation) to the no-CO2 standard approach.

The primary end point will be Time to Complete deairing as measured by intraoperative transesophageal echo while the secondary end point will be the incidence of clinical neurological events the day after the operation.

ELIGIBILITY:
Inclusion Criteria:

Isolated, Elective Aortic Valve Replacement or combined AVR and CABG

-

Exclusion Criteria:

* any other kind of operation
* Urgency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Time to Complete Deairing | Intraoperative
  Number of seconds since Declamping until no more air bubbles are visible on TEE Echo

SECONDARY OUTCOMES:
Neurological Events at Wake Up | The day after operation
  Either Convulsions, Transitory Ischemic Attack or Full Stroke

CONTACTS AND LOCATIONS:
Overall Officials: Luca Weltert, MD, Principal Investigator — European Hospital HEart Surgeon - Unicamillus Professor of Biostatistics
Locations (1):
- Cardiochirurgia European Hospital, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nyman J, Svenarud P, van der Linden J. Carbon dioxide de-airing in minimal invasive cardiac surgery, a new effective device. J Cardiothorac Surg. 2019 Jan 17;14(1):12. doi: 10.1186/s13019-018-0824-4. PMID 30654802
- [Background] Listewnik M, Kotfis K, Slozowski P, Mokrzycki K, Brykczynski M. The influence of carbon dioxide field flooding in mitral valve operations with cardiopulmonary bypass on S100ss level in blood plasma in the aging brain. Clin Interv Aging. 2018 Sep 25;13:1837-1845. doi: 10.2147/CIA.S177356. eCollection 2018. PMID 30288036
- [Background] Benedetto U, Caputo M, Guida G, Bucciarelli-Ducci C, Thai J, Bryan A, Angelini GD. Carbon Dioxide Insufflation During Cardiac Surgery: A Meta-analysis of Randomized Controlled Trials. Semin Thorac Cardiovasc Surg. 2017 Autumn;29(3):301-310. doi: 10.1053/j.semtcvs.2017.05.002. Epub 2017 May 23. PMID 29195572
- [Background] Ganguly G, Dixit V, Patrikar S, Venkatraman R, Gorthi SP, Tiwari N. Carbon dioxide insufflation and neurocognitive outcome of open heart surgery. Asian Cardiovasc Thorac Ann. 2015 Sep;23(7):774-80. doi: 10.1177/0218492315583562. Epub 2015 May 4. PMID 25939908
- [Background] Chatterjee S, Greenberg SB, Brown J, Murphy GS, Pearson PJ, Alexander JC. Simple technique to verify CO(2) diffusion with the CarbonAid device. Heart Surg Forum. 2012 Aug;15(4):E212-4. doi: 10.1532/HSF98.20121015. PMID 22917826
- [Background] Chaudhuri K, Storey E, Lee GA, Bailey M, Chan J, Rosenfeldt FL, Pick A, Negri J, Gooi J, Zimmet A, Esmore D, Merry C, Rowland M, Lin E, Marasco SF. Carbon dioxide insufflation in open-chamber cardiac surgery: a double-blind, randomized clinical trial of neurocognitive effects. J Thorac Cardiovasc Surg. 2012 Sep;144(3):646-653.e1. doi: 10.1016/j.jtcvs.2012.04.010. Epub 2012 May 12. PMID 22578685
- [Background] Al-Rashidi F, Landenhed M, Blomquist S, Hoglund P, Karlsson PA, Pierre L, Koul B. Comparison of the effectiveness and safety of a new de-airing technique with a standardized carbon dioxide insufflation technique in open left heart surgery: a randomized clinical trial. J Thorac Cardiovasc Surg. 2011 May;141(5):1128-33. doi: 10.1016/j.jtcvs.2010.07.013. Epub 2010 Sep 3. PMID 20817209
- [Background] Martens S, Neumann K, Sodemann C, Deschka H, Wimmer-Greinecker G, Moritz A. Carbon dioxide field flooding reduces neurologic impairment after open heart surgery. Ann Thorac Surg. 2008 Feb;85(2):543-7. doi: 10.1016/j.athoracsur.2007.08.047. PMID 18222261